CLINICAL TRIAL: NCT04980170
Title: Clindamycin Versus Amoxicillin With Clavulanic Acid in Prevention of Early Dental Implants Failure
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jordan University Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Hamdan, Oral and Maxillofacial surgery resident, Jordan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JordanUH
Record Dates: First submitted 2021-06-09; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Antibiotics Causing Adverse Effects in Therapeutic Use
Keywords: Effect of antiobiotic presctibed on early deental implant failure
MeSH Terms: interventions — Clindamycin; Amoxicillin; Clavulanic Acid; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clindamycin group (Experimental): Patients who take Clindamycin after Dental implants
  Interventions: Drug: Clindamycin 300 mg
- Amoxicillin With Clavulanic Acid group (Experimental): Patients who take Amoxicillin With Clavulanic Acid after Dental implants
  Interventions: Drug: Amoxicillin with Clavulanic Acid 635mg

INTERVENTIONS:
Drug: Clindamycin 300 mg — patients will be given clindamycin 300 mg twice daily for 5 days after dental implant
  Other Names: Clinacin
  Arms: clindamycin group
Drug: Amoxicillin with Clavulanic Acid 635mg — patients will be given Amoxicillin with Clavulanic Acid 635mg, three times daily for 5 days after dental implant
  Other Names: Augmentin
  Arms: Amoxicillin With Clavulanic Acid group

SUMMARY:
Among patients receiving dental implants, does the choice of antibiotics reduce the frequency of early implant failure ?

DETAILED DESCRIPTION:
The patients were selected in the implant assessment clinic from a population on the implant waiting list at the department of Maxillofacial surgery department , of Jordan University Hospital. Those consecutively assessed patients that complied with both the inclusion and the exclusion criteria and who had signed consent for participation in the study formed the study sample.

The following inclusion criteria were applied: • Presence of a partial edentulous or edentulous alveolar ridge. • Presence of a tooth or several teeth regarded as non-restorable with the intention of immediate implant placement. • Periodontally healthy remaining dentition. • Presence of a non-infected surgical site. • Presence of enough bone and soft tissue for the implant to be placed without additional augmentation procedures.

The following exclusion criteria were applied: • Patients with medical conditions that required antibiotic premedication such as prosthetic heart valve replacement, skeletal joint replacement, previous history of infective endocarditis and a history of rheumatic fever. • Patients with metabolic diseases such as type I or II diabetes mellitus. • Patients with past and present neoplastic disease. • Previous radiotherapy in the head and neck area. • Immunosuppressed patients. • Patients with blood coagulation impairment. • Patients with a history of systemic steroid medication or recent systemic antibiotic therapy. • Pregnant and lactating women • Patients with allergy to the antibiotic chosen Every patient that agreed to participate was randomly assigned to one of the following two groups: • First group - 625mg of AMOCLAN immediately postoperatively, three times a day for 5 days. • Secondl group - 600mg of CLINDAMYCIN immediately postoperatively, three times a day for 5 days. Consecutively treated patients received consecutive numbers correlating with the number of an envelope. This envelope contained either the 625mg Amoclan, or 600mg Clindamycin An independent person administered the antibiotic Neither the surgeon nor the patient knew which has been taken to ensure a double-blind approach One Professor in MaxFAx surgery was the operator One implant typr used: Blue Sky Bio, USA Implants were placed according to the manufacturers guidelines using standard surgical procedures. The local anaesthetic used was Articaine 4% with adrenaline 1 : 100,000.

Following adequate local anaesthesia, a mucoperiosteal flap was raised with or without one or two relieving incisions as determined by the local anatomy, including availability of bone, presence of neighbouring tooth roots and aesthetics. Osteotomies were then carried out under copious saline irrigation. Implants were then placed with a view to obtaining good primary stability. A decision was then made placing a cover screw and opting for a two stage approach . Closure of the surgical site with either resorbable or non-resorbable sutures was then performed ensuring tension free closure of the flaps.

The patient was personally instructed and handed out standardised forms on post-operative care. Patients were advised on the use of post-operative pain medication. To minimise the influence of independent variables, all patients were instructed to use paracetamol 500 mg tablets as required to a maximum of 4 g/day and Ibuprofen 400mg tablets to a maximum of 2000mg. Patients were advised to remain on a soft diet for the first post-operative week. Patients were instructed to use a chlorhexidine 0.2% mouthwash 4-5 times daily for the first postoperative week.

Recordings of osseointegration failure or success were recorded three months post-operatively or at 2nd stage surgery. Post-operative swelling was recorded on the 7th days.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a partial edentulous or edentulous alveolar ridge.
* Presence of a tooth or several teeth regarded as non-restorable with the intention of immediate implant placement.
* Periodontally healthy remaining dentition.
* Presence of a non-infected surgical site.
* Presence of enough bone and soft tissue for the implant to be placed without additional augmentation procedures.

  * Must be able to swallow tablets

Exclusion Criteria:

* Patients with medical conditions that required antibiotic premedication such as prosthetic heart valve replacement, skeletal joint replacement, previous history of infective endocarditis and a history of rheumatic fever.
* Patients with metabolic diseases such as type I or II diabetes mellitus.
* Patients with past and present neoplastic disease.
* Previous radiotherapy in the head and neck area.
* Immunosuppressed patients.
* Patients with blood coagulation impairment.
* Patients with a history of systemic steroid medication or recent systemic antibiotic therapy.
* Pregnant and lactating women
* Patients with allergy to the antibiotic chosen.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Early failure of osseointegration of dental implants | 3 months
  Failure of osseointegration is defined as having ANY ONE of the following during the first three months of implant placement.
  1. implant mobility: Measured using two metal instruments moving against each other.
  2. Acute surgical site infection: presence of erythema, swelling, pain, discharge at the site of implant.
  3. Radiographic Bone Loss >50% of implant length: measured using calibrated digital tool on peri-apical radiograph.
  4. Pain on function: measured using a verbal analogue scale (VAS). Patients were asked to describe the amount of pain they felt by giving a number from 0 to 10, where 0 represented not feeling any sort of pain and 10 represented the maximum pain they could imagine.

CONTACTS AND LOCATIONS:
Overall Officials: ASHRAF ABUKARAKI, PROFESSOR, Study Director — Jordan University Hospital
Locations (1):
- The University of Jordan Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared. But the final results of anonomysed individuals will be shared

REFERENCES:
- [Result] Malm MO, Jemt T, Stenport VF. Patient factors related to early implant failures in the edentulous jaw: A large retrospective case-control study. Clin Implant Dent Relat Res. 2021 Jun;23(3):466-476. doi: 10.1111/cid.13009. Epub 2021 May 17. PMID 33999522
- [Result] Malm MO, Jemt T, Stenport V. Early Implant Failures in Edentulous Patients: A Multivariable Regression Analysis of 4615 Consecutively Treated Jaws. A Retrospective Study. J Prosthodont. 2018 Dec;27(9):803-812. doi: 10.1111/jopr.12985. Epub 2018 Oct 29. PMID 30307086
- [Result] De Bruyn H, Raes S, Ostman PO, Cosyn J. Immediate loading in partially and completely edentulous jaws: a review of the literature with clinical guidelines. Periodontol 2000. 2014 Oct;66(1):153-87. doi: 10.1111/prd.12040. PMID 25123767
- [Result] Baqain ZH, Moqbel WY, Sawair FA. Early dental implant failure: risk factors. Br J Oral Maxillofac Surg. 2012 Apr;50(3):239-43. doi: 10.1016/j.bjoms.2011.04.074. Epub 2011 May 25. PMID 21612850